CLINICAL TRIAL: NCT06872164
Title: Onsite PTSD Treatment to Improve MOUD Outcomes: Open Pilot Trial of Stakeholder-engaged Adapted Cognitive Processing Therapy
Brief Title: Open Pilot Trial of Adapted Cognitive Processing Therapy for Comorbid PTSD and Opioid Use Disorder
Acronym: OPTIMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Teresa Lopez-Castro, Associate Professor, The City College of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 2025-16601; R61DA059032 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Opioid Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Cognitive Processing Therapy (Experimental): Participants will receive 4-18 sessions of telehealth-delivered Cognitive Processing Therapy (CPT) adapted for people who use syringe services programs. Participants will attend the 50-minute CPT sessions in a private space within the syringe services program.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT) is an evidence-based psychotherapy for PTSD that provides education and teaches skills to challenge the trauma-related beliefs that maintain PTSD symptoms. In this study, CPT has been adapted to include content on the relationship between substance use and PTSD and a focus on harm reduction.

SUMMARY:
The goal of this open pilot trial is to learn if an adapted version of Cognitive Processing Therapy (CPT), delivered through telehealth, can treat posttraumatic stress disorder (PTSD) in adults who use syringe services programs. The main questions it aims to answer are:

* Can the intervention be done in syringe services programs?
* Are syringe services program clients and staff open to the intervention?
* Can the intervention lower PTSD symptoms and help participants keep taking their medication for opioid use disorder (ex. Buprenorphine or methadone)?

Participants will:

* Attend 4-18 tele-delivered CPT sessions at the syringe services program
* Complete between-session CPT practice with the support of SSP-based "coaches"
* Meet with research staff monthly to complete surveys of their PTSD symptoms, drug use, and mental health

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Regular syringe services program attendance (ex. at least 4 visits in the past month)
* Meeting DSM-5 opioid use disorder criteria
* Having been prescribed a medication for opioid use disorder in the past 30 days at the time of screening
* Criterion A event as measured by the Life Events Checklist for DSM-5 (LEC-5)
* PTSD symptoms at the level of a PTSD diagnosis as evidenced by a score of 31 or greater on the PTSD Checklist for DSM-5 (PCL-5)
* Ability to understand English
* Consent to have assessment interviews audio recorded and teletherapy sessions video recorded for research purposes
* Ability to provide informed consent

Exclusion Criteria:

* High risk for suicidal thoughts and/or behaviors that would make participation dangerous, as measured by the Columbia Suicide Severity Rating Scale Lifetime-Recent Screen
* Meeting DSM-5 criteria for a current psychotic or bipolar disorder.
* Cognitive impairment liable to interfere with completion of study procedures
* Currently receiving trauma-focused psychotherapy (i.e. Prolonged Exposure, Cognitive Processing Therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Eligible Participants | Baseline
  Proportion of persons eligible to enroll in the study of all possible SSP clients approached during 6-month recruitment period. Assessed using count data of individuals failing screen.
Proportion of Eligible Participants who Enroll | Week 1
  Proportion of all eligible persons who enroll. Assessed using count data of individuals consented.
Mean Number of Intervention Sessions Attended | Up to Week 12
  Mean number of teletherapy sessions attended by enrolled participants. Assessed using count data of session attendance.
Proportion of Study Visits Completed by Enrolled Participants | Week 12
  Proportion of study visits completed by enrolled participants. Assessed using count data of study visit attendance.
Proportion of Participants With at Least one SSP-based Coach Encounter | Week 12
  Proportion of participants who have attended at least one teletherapy sessions and have had at least one SSP-based coach encounters.
Participant-rated Client Satisfaction Questionnaire Score | Week 12
  8-item, participant-rated assessment of satisfaction with intervention. Total score is the sum of responses and ranges from 8 to 32. Higher scores indicate greater client satisfaction and treatment acceptability.
Therapist & Coach-Rated Feasibility of Intervention Measure Score | Week 12
  Four-item, clinician-rated assessment of the feasibility of the intervention. Each item is rated on a scale from 1 (Completely disagree) to 5 (Completely agree); the total score is the sum of responses and ranges from 4-20. Higher scores indicate greater clinician-rated feasibility.
Therapist & Coach-Rated Acceptability of Intervention Measure Score | Week 12
  Four-item, clinician-rated assessment of the acceptability of the intervention. Each item is rated on a scale from 1 (Completely disagree) to 5 (Completely agree); the total score is the sum of responses and ranges from 4-20. Higher scores indicate greater clinician-rated acceptability.
Therapist & Coach-Rated Intervention Appropriateness Measure Score | Week 12
  Four-item, clinician-rated assessment of whether the intervention is appropriate for the setting and target population. Each item is rated on a scale from 1 (Completely disagree) to 5 (Completely agree); the total score is the sum of responses and ranges from 4-20. Higher scores indicate greater clinician-rated appropriateness.

SECONDARY OUTCOMES:
Change From Baseline in PCL-5 Total Score | Baseline and Week 12
  The PCL-5 has 20 items assessing PTSD symptom severity. Total scores range from 0-80 with higher scores indicating more severe PTSD symptoms. The score at baseline will be subtracted from the score at week 12.
Changes from baseline in self-reported past 30-day use of prescribed MOUD | Baseline and Week 12
  Number of self-reported days in the past 30 days in which prescribed MOUD was taken. The number at baseline will be subtracted from the number at week 12.
Changes from baseline in self-reported days of nonprescribed opioids | Baseline and Week 12
  Number of self-reported days of nonprescribed opioids in past 30 days using the Drug Use section of the Addiction Severity Index. The number at baseline will be subtracted from the number at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lopez-Castro, PhD, Principal Investigator — The City College of New York, CUNY; Aaron D Fox, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- OnPoint, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected, deidentified individual patient data from enrolled participants of the open trial will be shared. Final datasets will include self-reported psychosocial, demographic, and behavioral data from interviews, and urine toxicology data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available upon completion of the multi-site trial (2029).
Access Criteria: Given that deidentified data will contain sensitive information, it will be archived at the National Addiction & HIV Data Archive Program NAHDAP, a controlled-access repository. Data will be findable via NAHDAP's persistent unique identifiers.